CLINICAL TRIAL: NCT00005790
Title: Perfusion Magnetic Resonance Imaging of Brain Tumors: Correlation With Indicators of Angiogenesis
Brief Title: Perfusion Magnetic Resonance Imaging in Measuring the Growth of Blood Vessels in Newly Diagnosed Brain Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to accrue subjects.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: NU 95C1; NU-95C1; NCI-G00-1738
Record Dates: First submitted 2000-06-02; First posted 2004-06-09 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult brain stem glioma; adult ependymoma; adult craniopharyngioma; adult medulloblastoma; adult meningioma; adult glioblastoma; adult oligodendroglioma; adult anaplastic astrocytoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult pineal parenchymal tumor; adult central nervous system germ cell tumor; adult pilocytic astrocytoma; adult subependymoma; adult diffuse astrocytoma; adult ependymoblastoma; adult pineocytoma; adult pineoblastoma; adult meningeal hemangiopericytoma; adult choroid plexus tumor; adult grade III meningioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Ependymoma; Craniopharyngioma; Medulloblastoma; Meningioma; Glioblastoma; Oligodendroglioma; Astrocytoma; Glioma; Pinealoma; Glioma, Subependymal; Neuroectodermal Tumors, Primitive; Choroid Plexus Neoplasms; Gliosarcoma | interventions — Biopsy; Magnetic Resonance Spectroscopy; Gadolinium DTPA

INTERVENTIONS:
Other: laboratory biomarker analysis
Procedure: biopsy
Procedure: magnetic resonance imaging
Radiation: gadopentetate dimeglumine

SUMMARY:
RATIONALE: Perfusion magnetic resonance imaging may be an effective method of measuring the growth of blood vessels in brain tumors. These measurements may help doctors better diagnose and treat brain tumors.

PURPOSE: Pilot study to determine the effectiveness of perfusion magnetic resonance imaging in measuring the growth of blood vessels in newly diagnosed brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Correlate the findings of perfusion magnetic resonance imaging with known tissue and serum markers of angiogenesis in patients with newly diagnosed surgically resectable brain tumors.

OUTLINE: Patients undergo perfusion magnetic resonance imaging (MRI) scanning with contrast in conjunction with preoperative conventional MRI scanning with contrast. Patients receive gadopentetate dimeglumine IV over 5 seconds prior to perfusion MRI. Gadopentetate dimeglumine is administered at a slower rate prior to conventional MRI. Patients undergo blood draw to determine urokinase type plasminogen activator levels. After completion of perfusion and conventional MRI scanning, brain tumor tissue samples are obtained during surgical resection to determine tumor grade and type and urokinase type plasminogen activator and basic fibroblast growth factor levels. If CSF removal is required during surgery, then CSF samples are collected to determine urokinase type plasminogen activator and basic fibroblast growth factor levels.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed surgically resectable brain tumor

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Able to tolerate gadopentetate dimeglumine contrast Medically stable

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1996-04; Primary Completion 1999-05; Study Completion 1999-05

CONTACTS AND LOCATIONS:
Overall Officials: Hunt H. Batjer, MD, Study Chair — Robert H. Lurie Cancer Center